CLINICAL TRIAL: NCT03381703
Title: A Phase I Study to Investigate the Absorption, Metabolism, and Excretion and the Absolute Bioavailability of YH12852 in Healthy Male Subjects
Brief Title: Investigation of the Absorption, Metabolism, and Excretion and the Absolute Bioavailability of YH12852
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YH12852-103(I)
Record Dates: First submitted 2017-10-29; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2016-05

CONDITIONS: Constipation
Keywords: Accelerated Mass Spectrometry; Microtracer; Microdose; hAME; Absolute bioavailability
MeSH Terms: conditions — Constipation | interventions — YH12852

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Investigate the absorption, metabolism, and excretion of YH12852
  Interventions: Drug: YH12852; Drug: 14C-labeled YH12852
- Part 2 (Experimental): Investigate the absolute bioavailability of YH12852
  Interventions: Drug: YH12852; Drug: 14C-labeled YH12852

INTERVENTIONS:
Drug: YH12852 — YH12852 administration
Drug: 14C-labeled YH12852 — 14C-labeled YH12852 administration

SUMMARY:
This study investigates the absorption, metabolism, and excretion and the absolute bioavailability of YH12852 in healthy male subjects

DETAILED DESCRIPTION:
Part 1 : Investigate the absorption metabolism, and excretion of YH12852 after single oral administration of YH12852 and 14C-labeled YH12852.

Part 2

: Investigate the absolute bioavailability of YH12852 after single oral administration of YH12852 followed by a single i.v. administration of 14C-labeled YH12852.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agreed to voluntarily participate in this study and comply with all the study requirements by signing informed consent form after being informed of the nature of this study and understanding all aspects of this study
* Healthy adult, 19 - 55 of age (inclusive)
* Subjects weighing over 55 kg (inclusive) with BMI between 18 and 25 (inclusive) at screening visit
* Subjects with no clinically significant abnormal findings as determined by physical examination, ECG, medical history, or clinical laboratory test results

Exclusion Criteria:

* History of clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorder
* Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug
* History of (or suspected at screening visit) disease listed below Myocardial infarction Cerebral infarction/Stroke Arrythmia that need medical treatment Unstable angina Pulmonary hypertension
* Subjects who are positive for Hepatitis B, Hepatitis C, and HIV
* History of relevant allergy/hypersensitivity
* Subjects who took prescribed medications within 14 days or over-the-counter (OTC) medications within 7 days prior to the first dose of the study drug
* Subjects who have been consuming over 21 unit(1 unit = 10 g of alcohol) per week of alcohol prior to the study initiation or who is not able to stop consuming alcohol throughout the hospitalization period
* Subjects who consumed products listed below within 2 days prior to the first dose of the study drug or who is not able to stop consuming products listed below until the last site visit Foods and/or beverages containing grapefruit Products containing caffeine (Coffee, tea, chocolate, caffeine-containing soft drinks)
* Subject who is not willing to use contraception throughout the study
* Subjects who have smoked over 10 cigarettes until 3 months prior to the study initiation or who is not able to stop smoking throughout the hospitalization period
* Subjects who have donated whole blood within 2 months or blood component within 1 month or received blood transfusion within 1 month of participating in this study
* Administration of any investigational products within 3 months from the first dose of the study drug
* Subject who's serum prolactin is over 3-fold higher than the upper limit of normal range
* Subject who judged not eligible for study participation by investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Total radioactivity | 0 - 288 hours (post-dose)
  Total radioactivity recovered
Cmax of YH12852 | 0(pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288 hours (post-dose)
  Peak concentration of YH12852
AUClast of YH12852 | 0(pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288 hours (post-dose)
  Area under the concentration-time curve from time 0 to the last measurable time of YH12852
Fpo of YH12852 | 0(pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288 hours (post-dose)
  Oral bioavailability of YH12852

SECONDARY OUTCOMES:
Aef of YH12852 | 0 - 288 hours (post-dose)
  Amount excreted in feces of YH12852
Aeu of YH12852 | 0 - 288 hours (post-dose)
  Amount excreted in urine of YH12852

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, MD., PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided